CLINICAL TRIAL: NCT03667937
Title: Effectiveness of a Hydrophobic Dressing for Microorganisms' Colonization and Infection Control of Vascular Ulcers: An Open, Controlled, Randomized Study, With Blinded Endpoint (PROBE Trial): CUCO-UV Study
Brief Title: Effectiveness of a Hydrophobic Dressing for Microorganisms' Colonization and Infection Control of Vascular Ulcers
Acronym: CUCO-UV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaga (Other)
Collaborators: BSN Medical GmbH (Industry); Andalusian Health Service (Other Government)
Responsible Party: Principal Investigator, JOSE MIGUEL MORALES ASENCIO, Head of the Department of Nursing. Professor of Research and Evidence Based Health Care, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUCO-UV
Record Dates: First submitted 2018-05-24; First posted 2018-09-12 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Venous Leg Ulcer; Bacterial Infections; Chronic Ulcer of Skin of Lower Limb Nos
Keywords: Venous Ulcer; Leg Injuries; Bacterial Infections
MeSH Terms: conditions — Varicose Ulcer; Bacterial Infections; Leg Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CUTIMED (Experimental): After an initial culture to determine the bacterial load by smear, we will proceed to the cure of the ulcer by washing the area with physiological saline solution and to mechanical debridement, if necessary, to apply the CUTIMED dressing. It will be covered with a secondary gauze dressing and a double compression bandage with a normal crepe bandage.
  If the wound exudate decreases, or the removal of the dressing is difficult, it will be changed to CUTIMED gel; in case of abundant exudate, the use of alginate without silver will be allowed for the treatment, because it is neutral with the bacterial load, placed on the CUTIMED dressing.
  Primary and secondary end-points will be measured at baseline and at 4, 8 and 12 weeks, except quality of life (only baseline and at 12 weeks).
  Interventions: Combination Product: CUTIMED
- AQUACEL silver (Active Comparator): After an initial culture to determine the bacterial load by smear, we will proceed to the cure of the ulcer by washing the area with physiological saline solution and to mechanical debridement, if necessary, to apply Aquacel-Ag. It will be covered with a secondary gauze dressing and a double compression bandage with a normal crepe bandage.
  Primary and secondary end-points will be measured at baseline and at 4, 8 and 12 weeks, except quality of life (only baseline and at 12 weeks).
  Interventions: Other: AQUACEL silver

INTERVENTIONS:
Combination Product: CUTIMED — Hydrophobic Dressing
  Arms: CUTIMED
Other: AQUACEL silver — Silver Dressing
  Arms: AQUACEL silver

SUMMARY:
This study will determine the effectiveness of CUTIMED® hydrophobic dressings against AQUACEL® silver dressings in bacterial colonization of vascular ulcers.

DETAILED DESCRIPTION:
Chronic wounds with torpid evolution are a real challenge for health services today. In the case of venous ulcers, it is estimated that more than 80% of these wounds may be colonized or infected by bacteria, which is associated with its chronification by delaying the healing process.

The most widespread therapeutic strategy in routine clinical practice is the use of silver dressings, due to its high antimicrobial power, although the effectiveness of these in venous ulcers is not supported by solid evidence. In addition, there are some uncertainties about the possible adverse effects of systemic absorption of silver molecules, as well as bacterial resistance to silver and the high cost associated with prolonged treatments.

In this sense, a novel method to deal with this problem is the use of dressings with high hydrophobic power, such as CUTIMED®.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with chronic venous vascular ulcer located in lower limbs with signs of critical colonization, according to the criteria of Lazareth and Moore, which imply the presence of at least 3 of the following five:

1. Severe pain during dressing change
2. Perilesional edema.
3. Local edema.
4. Unpleasant smell.
5. Abundant pus
6. Microbial colonization higher than 100000 CFUs

Exclusion Criteria:

* Patients younger than 18 years old.
* Venous ulcer with signs of infection which requires antibiotic therapy
* Venous ulcers that do not meet Lazareth and Moore criteria
* Arterial ulcers.
* Patients with type I or type II diabetes.
* Patients with immunosuppression of any etiology or in immunosuppressive treatment or with NSAIDs.
* Patients with rheumatoid arthritis in the acute phase.
* Patients with dermatitis prior to the appearance of the ulcer.
* Patients with neuropathy or lack of sensitivity of any etiology.
* Patients who, for local or systemic clinical reasons, will need to initiate antibiotic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Microorganisms' Colonization Level | Change from baseline, at 4, 8 and 12 weeks
  Evaluated by Reverse Transcription Polymerase Chain Reaction (RT-PCR) identification technique and quantified in colony forming units (CFU) and in ng of bacterial DNA per μL of vascular ulcer exudate.

SECONDARY OUTCOMES:
Pain due to the wound | Change from baseline at 4, 8 and 12 weeks
  Measured with tha Visual Analogue Scale (VAS): Minimum score=1; Maximum score=10.
Wound size (wound reduction percentage) | Baseline, 4, 8 and 12 weeks
  It will be evaluated by planimetry with PictZar 7.5 software
Healing time | Change from baseline at 4, 8 and 12 weeks
  This outcome will be measure by number of days until healing
Complete wound healing (Resvech 2.0 score) | Change from baseline at 4, 8 and 12 weeks
  Complete healing will be considered with a 0 score in the fourth dimension of the Resvech 2.0 scale
Patient quality of life | Change from baseline at 12 weeks
  Measured with Charing Cross Venous Ulcer Questionnaire (CCVUQ), in its Spanish version. The CCVUQ is composed of 22 items that determine four important dimensions for health: the social function, domestic activities, the aesthetic dimension and the emotional state. Each item should be assessed using a Likert scale with a punctuation from 1 to 5. In their interpretation, lower scores indicate a better quality of life.
Adverse Events | Change from baseline at 4, 8 and 12 weeks
  Adverse events related with the treatment, referred by patients, caregivers or health professionals

OTHER OUTCOMES:
Wound healing evolution | Baseline, 4, 8 and 12 weeks
  Measured with "Resultados esperados de la valoración y evolución de la cicatrización de las heridas crónicas" (Expected results of chronic wound healing assessment and evolution), RESVECH 2.0 scale. The punctuation varies forn 0 to 35, with 6 subscales: Wound size, Depth/affected tissues, Borders, Type of tissue in the wound bed, Type of exudate and Infection/inflammation

CONTACTS AND LOCATIONS:
Overall Officials: José Miguel Morales Asencio, PhD, Principal Investigator — University of Malaga
Locations (1):
- University of Málaga, Málaga, Spain

REFERENCES:
- [Background] Gonzalez de la Torre H, Quintana-Lorenzo ML, Perdomo-Perez E, Verdu J. Correlation between health-related quality of life and venous leg ulcer's severity and characteristics: a cross-sectional study. Int Wound J. 2017 Apr;14(2):360-368. doi: 10.1111/iwj.12610. Epub 2016 Apr 25. PMID 27112627
- [Background] Hansson L, Hedner T, Dahlof B. Prospective randomized open blinded end-point (PROBE) study. A novel design for intervention trials. Prospective Randomized Open Blinded End-Point. Blood Press. 1992 Aug;1(2):113-9. doi: 10.3109/08037059209077502. PMID 1366259
- [Background] Lazareth I, Ourabah Z, Senet P, Cartier H, Sauvadet A, Bohbot S. Evaluation of a new silver foam dressing in patients with critically colonised venous leg ulcers. J Wound Care. 2007 Mar;16(3):129-32. doi: 10.12968/jowc.2007.16.3.27015. PMID 17385590
- [Background] Moore K, Hall V, Paull A, Morris T, Brown S, McCulloch D, Richardson MC, Harding KG. Surface bacteriology of venous leg ulcers and healing outcome. J Clin Pathol. 2010 Sep;63(9):830-4. doi: 10.1136/jcp.2010.077032. Epub 2010 Jul 29. PMID 20671048
- [Background] Moore MF. Prospective, Descriptive Study of Critically Colonized Venous Leg Ulcers Managed With Silver Containing Absorbent Dressings and Compression. J Am Coll Clin Wound Spec. 2014 Sep 16;5(2):36-9. doi: 10.1016/j.jccw.2014.08.002. eCollection 2013 Aug. PMID 26199888
- [Background] Pugliese DJ. Infection in Venous Leg Ulcers: Considerations for Optimal Management in the Elderly. Drugs Aging. 2016 Feb;33(2):87-96. doi: 10.1007/s40266-016-0343-8. PMID 26833351
- [Background] Totty JP, Bua N, Smith GE, Harwood AE, Carradice D, Wallace T, Chetter IC. Dialkylcarbamoyl chloride (DACC)-coated dressings in the management and prevention of wound infection: a systematic review. J Wound Care. 2017 Mar 2;26(3):107-114. doi: 10.12968/jowc.2017.26.3.107. PMID 28277989
- [Background] Wendelken ME, Berg WT, Lichtenstein P, Markowitz L, Comfort C, Alvarez OM. Wounds measured from digital photographs using photodigital planimetry software: validation and rater reliability. Wounds. 2011 Sep;23(9):267-75. PMID 25879267
- [Background] González-Consuegra, R.V., Verdú, J., 2010. Proceso de adaptación al castellano del Charing Cross Venous Ulcer Questionnaire (CCVUQ) para medir la calidad de vida relacionada con la salud en pacientes con úlceras venosas. Gerokomos 21, 80-87